CLINICAL TRIAL: NCT05057702
Title: A Pilot Feasibility and Efficacy (Phase 2) Trial of Real Time Drug Screening and Genomic Testing to Determine an Individualized Treatment Plan in Children and Young Adults With Relapsed Medulloblastoma and Ependymoma
Brief Title: Individualized Treatment Plan in Children and Young Adults With Relapsed Medulloblastoma and Ependymoma
Acronym: PNOC027
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Washington University School of Medicine (Other); St. Baldrick's Foundation (Other); Ashion Analytics (Unknown); University of Washington (Other); Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 21083; NCI-2021-09726 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Medulloblastoma; Medulloblastoma, Childhood; Medulloblastoma Recurrent; Ependymoma; Ependymoma Malignant; Ependymoma of Brain
Keywords: Individualized Treatment Plan; Genetic Screening; Screening
MeSH Terms: conditions — Medulloblastoma; Ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized Treatment Recommendation (Pilot Phase) (Experimental): Participants will receive an individualized treatment recommendation including a combination of up to four FDA-approved drugs within 21 business days of tissue acquisition using the results of real-time high-throughput drug screening, whole exome sequencing (WES), and RNA sequencing.
  Interventions: Other: Specialized Tumor Board Treatment Plan; Other: Combinations
- Individualized Treatment Recommendation (Efficacy Phase) (Experimental): Participants will receive an individualized treatment recommendation including a combination of up to four FDA-approved drugs within 21 business days of tissue acquisition using the results of real-time high-throughput drug screening, whole exome sequencing (WES), and RNA sequencing.
  Interventions: Other: Specialized Tumor Board Treatment Plan; Other: Combinations

INTERVENTIONS:
Other: Specialized Tumor Board Treatment Plan — Specialized Treatment Plan of up to four FDA approved drugs based on participant's screening results will be assigned by PNOC specialized tumor board
  Other Names: Individualized Treatment Plan; Specialized Treatment Plan
Other: Combinations — Specialized Treatment Plan of up to four FDA approved drugs based on participant's screening results will be assigned by PNOC specialized tumor board
  Other Names: Multiple Treatments Physician Discretion

SUMMARY:
The current study will use a new treatment approach based on the molecular characteristics of each participant's tumor. The study will test the feasibility in the pilot phase of performing real-time drug screening on tissue taken during surgery in patients with relapsed medulloblastoma or ependymoma and of having a specialized tumor board assign a treatment plan based on the results of this screening and genomic sequencing. The aim of this trial is to allow every child and young adult with relapsed medulloblastoma and ependymoma to receive the most effective and least toxic therapies currently available and will pave the way for improved understanding and treatment of these tumors in the future. Moreover, if successful, it could serve as a paradigm for personalized medicine programs for other types of cancer.

DETAILED DESCRIPTION:
This is a multi-center pilot trial within the Pacific Pediatric Neuro-Oncology Consortium (PNOC). Relapsed participants will receive an individualized treatment recommendation including up to four FDA-approved drugs based on the results of real-time high-throughput drug screening, whole exome sequencing (WES), and RNA sequencing.

PRIMARY OBJECTIVE:

For pilot phase (CLOSED TO ENROLLMENT):

I. To determine the feasibility of using the results of real-time in vitro drug screening, whole exome sequencing, and RNA sequencing of participant-derived specimens to guide treatment recommendations by a specialized tumor board, in a clinically actionable timeframe, for children and young adults with recurrent medulloblastoma or ependymoma

For efficacy phase:

II. To determine the progression-free survival (PFS) in children and young adults with relapsed medulloblastoma and ependymoma who received the specialized tumor board recommendation and compare to historical cohorts.

SECONDARY OBJECTIVE:

For pilot (CLOSED TO ENROLLMENT) and efficacy phases:

I. To determine the safety and describe the toxicity of treating children and young adults with relapsed medulloblastoma and ependymoma according to a specialized tumor board recommended treatment plan.

EXPLORATORY OBJECTIVES:

Pilot Phase (CLOSED TO ENROLLMENT):

I. To estimate the objective response rate, progression free survival at 6 months (PFS-6) and overall survival (OS) of relapsed medulloblastoma in children and young adults treated with an individualized treatment regimen.

II. To assess Quality of Life (QOL) measures in participants with relapsed medulloblastoma treated with an individualized regimen.

III. To archive tumor and normal DNA from each participant along with serial blood draw following therapies as biospecimens for later studies to determine whether cfDNA sequences in the participant's blood serve as biomarkers of tumor burden, response to therapy, or development of drug resistance.

Efficacy Phase:

I. To determine the overall survival (OS) and objective response rate (ORR) in children and young adults with relapsed medulloblastoma and ependymoma who received the specialized tumor board recommendation and compare to historical cohorts.

II. To generate PDX models of relapsed medulloblastoma and ependymoma to facilitate future in vivo testing of therapeutic agents.

III. To assess the correlation between available genomic data (WES and RNAseq) and patient outcomes, evaluating its potential complementary role in guiding therapeutic decisions alongside the primary drug screening approach.

IV. To archive tumor and normal DNA from each participant along with serial blood draw following therapies as biospecimens for later studies to determine whether cell free DNA (cfDNA) sequences in the participant's blood serve as biomarkers of tumor burden, response to therapy, or development of drug resistance.

V. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures in the context of race ethnicity and other health related social risks.

VI. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks.

Participants were initially enrolled in a pilot phase (CLOSED TO ENROLLMENT), and additional participants will be enrolled in the efficacy phase. Participants may continue treatment as tolerated for up to two years or until disease progression. After two years, patients may be eligible to continue therapy if they are experiencing clinical benefits, have disease control, and it is deemed appropriate to do so by their physician. Participants will be followed until progression, death, or up to 5 years from start of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have recurrent medulloblastoma or recurrent ependymoma previously histologically confirmed. Participants must be experiencing their first or second relapse to be eligible.
2. Participants must have surgically accessible disease.
3. Prior Therapy:

   1. The participant must have received at least one prior therapy at the time of initial diagnosis.
   2. Relapsed medulloblastoma or relapsed ependymoma are eligible.
   3. Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and would be eligible for surgical resection per institutional guidelines

      * Participants must have received last chemotherapy or biologic agent at least 7 days prior to registration.
      * Monoclonal antibody treatment: > 21 days prior to registration.
      * Bevacizumab participants must have received last dose > 21 days prior to study registration
4. Participant must be a candidate for surgical resection or biopsy with anticipated ability to obtain the minimum tissue requirements for study.
5. Radiation - Participants must have:

   1. Had their last fraction of local irradiation to primary tumor >= 12 weeks prior to registration.
   2. Had their last fraction of craniospinal irradiation or total body irradiation >= 12 weeks prior to registration
   3. At least 14 days after local palliative radiation (small-port)
6. Age >=12 months to <= 39 years of age.
7. Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants <= 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
8. Corticosteroids: Participants who are receiving dexamethasone or equivalent must be on a stable or decreasing dose for at least 1 week prior to registration.
9. Organ Function Requirements (within 7 days prior to study registration)

   1. Adequate Bone Marrow Function Defined as:

      * Peripheral absolute neutrophil count (ANC) >= 750/mm^3
      * Platelet count >= 75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
      * Hemoglobin >= 8 g/dl.
   2. Adequate Renal Function Defined as:

      * Creatinine clearance or radioisotope GFR >= 70 milliliter/minute (mL/min) /1.73 m^2 or
      * A serum creatinine based on age/sex as follows:

      Age / Maximum Serum Creatinine (mg/dL) Male / Maximum Serum Creatinine (mg/dL) Female.
      * 1 to < 2 years / 0.6 / 0.6.
      * 2 to < 6 years / 0.8 / 0.8.
      * 6 to < 10 years / 1 / 1.
      * 10 to < 13 years / 1.2 / 1.2.
      * 13 to < 16 years / 1.5 / 1.4.
      * >= 16 years / 1.7 / 1.4.
      * - The threshold creatinine values in this table were derived from the Schwartz formula for estimating Glomerular filtration rate (GFR) utilizing child length and stature data published by the Center for Disease Control (CDC) (Schwartz GJ and Gauthier B 1985).
   3. Adequate Liver Function Defined as:

      * Total Bilirubin <= 1.5 x upper limit of normal (ULN) for age; in presence of Gilbert's syndrome, total bilirubin < 3 x ULN or direct bilirubin < 1.5 x ULN.
      * Alanine aminotransferase (ALT) <= 3x ULN.
      * Aspartate aminotransferase (AST) <= 3x ULN.
10. The effects of the agents used in this study on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of therapy administration. Should a woman become pregnant or suspect pregnancy while participating in this study, the treating physician should be informed immediately.
11. Adequate neurologic function defined as participants with seizure disorder may be enrolled if seizures are well controlled. Participants on non-enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drug.
12. Participants must enroll on the Protocol for Children and Young Adults Diagnosed with a Central Nervous System (CNS) Tumor to Assess Cognitive, Quality of Life (QOL), and Comprehensive Effects of Therapies (PNOC COMP) study if PNOC COMP is open to accrual at the enrolling institution
13. A legal parent/guardian or participant must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.

Exclusion Criteria:

1. Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Participants who are receiving any other investigational agents.
3. Participants must be at least 7 days since the completion of therapy with a biologic or small molecule agent. For any agent with known adverse events that can occur beyond 7 days after administration, the period prior to enrollment must be beyond the time during which adverse events are known to occur. Such participants should also be discussed with study chairs.
4. Participants who are currently taking any anti-cancer direct therapy. Steroids are not considered anti-cancer therapy.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
6. Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required prior to start of therapy.
7. Participants must not receive any tumor-directed therapy after enrollment, except for surgical resection/ biopsy.

Important note: The eligibility criteria listed above are interpreted literally and cannot be waived.

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants for whom treatment recommendations are fully completed within 21 business days of tissue collection based on drug screening (Pilot Phase) | Up to 21 days
  Time to tissue collection will be used to determine the feasibility of using the results of real-time in vitro drug screening, WES and RNAseq of participant-derived specimens to guide treatment recommendations by a specialized tumor board, in a clinically-actionable timeframe, for children and young adults with recurrent medulloblastoma. Participants are expected to receive treatment plan within 21 business days
Percentage of participants with treatment recommendations within 21 business days (Pilot Phase) | Up to 21 days
  Time to tissue collection will be used to determine the feasibility of using the results of real-time in vitro drug screening, WES and RNAseq of participant-derived specimens to guide treatment recommendations by a specialized tumor board, in a clinically-actionable timeframe, for children and young adults with recurrent medulloblastoma. Participants are expected to receive treatment plan within 21 business days
Number of participants without adequate tissue | Up to 21 days
  The number of consented participants who do not have adequate tissue collection will be used to determine the feasibility.
Median Time from tissue collection to issued treatment plan from the specialized tumor board (Pilot Phase) | Up to 21 days
  Time to tissue collection will be used to determine the feasibility of using the results of real-time in vitro drug screening, WES and RNAseq of participant-derived specimens to guide treatment recommendations by a specialized tumor board, in a clinically-actionable timeframe, for children and young adults with recurrent medulloblastoma. Participants are expected to receive treatment plan within 21 business days
Median Progression-free survival (PFS) (Efficacy Phase) | Up to 5 years
  The median months from the time of surgery for this recurrence to the first evidence of progression or death, using PFS at 10 months (PFS10) for the relapsed medulloblastoma cohort and PFS at 17 months for the relapsed ependymoma cohort (Arm B).

SECONDARY OUTCOMES:
Proportion of participants with Adverse Events | Up to 2 years
  Proportion of participants with grade 3 or higher toxicities classified according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events and clinically significant laboratory abnormalities (meeting Grade 3 or higher criteria will be summarized by maximum grade and relationship to study drug(s).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Robert Wechsler-Reya, PhD, Study Chair — Columbia University; Margaret Shatara, MD, Study Chair — Washington University School of Medicine; Megan Paul, MD, Study Chair — Rady Children's Hospital; Lindsay Kilburn, MD, Study Chair — Children's National Research Institute
Locations (8):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - St. Louis Children's Hospital / Washington University in St. Louis, St Louis, Missouri
  - New York University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol